CLINICAL TRIAL: NCT03453138
Title: The Comparison of Protector LMA and Endotracheal Tube in Patients Undergoing Laparoscopic Cholecystectomy Under General Anesthesia A Randomize Controlled Trial
Brief Title: Usage of LMA Protector on Patients Who Undergo Laparoscopic Surgery
Acronym: LMAP-LS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayse Zeynep Turan, Principal Investigator, Derince Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DerinceTRH-01
Record Dates: First submitted 2018-01-29; First posted 2018-03-05 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Laryngeal Mask Airway
Keywords: laryngel mask airway; laparoscopic surgery
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LMA Protector Group (Experimental): LMA Protector will be inserted by a blind researcher after standart anesthesia induction. The view of the larynx will be assessed using fiberoptic grading scale
  Interventions: Device: LMA Protector
- Tracheal Intubation Group (Experimental): Patients will be intubated after standart anesthesia induction and we will record heamodynamic variables. including mean blood pressure and heart rate
  Interventions: Device: Tracheal Intubation

INTERVENTIONS:
Device: LMA Protector — LMA Protector will be inserted by a blind researcher after standart anesthesia induction. The view of the larynx will be assessed using fiberoptic grading scale
  Arms: LMA Protector Group
Device: Tracheal Intubation — tracheal intubation will be perform after standart anaesthetic induction and heamodynamic variables including blood pressure heart rate and possible complications will be observed
  Arms: Tracheal Intubation Group

SUMMARY:
LMA Protector is a recently developed second generation laryngeal mask several kinds of different laryngeal masks were used for the airway management during laparoscopic surgeries. However there is a lack of knowledge for the use of LMA Protector during laparoscopic surgery .In this study researchers aim to determine the effectivity of LMA Protector and plan to analyse the orofaryngeal cuff pressure and fiberoptic grading scale measurements .

DETAILED DESCRIPTION:
Tracheal intubation may have more complications than laryngeal masks. In this study researchers aim to determine the effectivity of LMA Protector and on the otherside the heamodynamic variables and the complication rates between tracheal ıntubation and laryngeal mask insertion will be compared.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I-III patients
* Patients undergo laparoscopic surgeries
* Laparoscopic surgeries duration of less than 2 hours

Exclusion Criteria:

* Difficult intubation history
* BMI>35
* Open cholesistectomies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2017-12-26 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Ventilatory efficiency pressures for the LMA Protector | Intraoperative
  Oropharyngeal pressure leak test, the peak airway pressures will be determined

SECONDARY OUTCOMES:
Feasibility of LMA Protector | Intraoperative
  The grading of fiberoptic view of larynx through the LMA Protector
Ease of insertion of LMA Protector | Intraoperative
  Each attemption to insert LMA will be record.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Yılmaz, MD, Principal Investigator — Derince Research and Training Hospital
Locations (1):
- Derince Research and Training Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
the reason is not to cause bias between the researchers

REFERENCES:
- [Background] Singh K, Gurha P. Comparative evaluation of Ambu AuraGain with ProSeal laryngeal mask airway in patients undergoing laparoscopic cholecystectomy. Indian J Anaesth. 2017 Jun;61(6):469-474. doi: 10.4103/ija.IJA_163_17. PMID 28655951
- [Background] Park SY, Rim JC, Kim H, Lee JH, Chung CJ. Comparison of i-gel(R) and LMA Supreme(R) during laparoscopic cholecystectomy. Korean J Anesthesiol. 2015 Oct;68(5):455-61. doi: 10.4097/kjae.2015.68.5.455. Epub 2015 Sep 30. PMID 26495055